CLINICAL TRIAL: NCT01273441
Title: Phase 4, Prospective, Randomized and Comparative Study Comparing Sequential and Concomitant Therapy for Helicobacter Pylori Eradication in Routine Clinical Practice
Brief Title: Study Comparing Sequential and Concomitant Therapy for Helicobacter Pylori Eradication in Routine Clinical Practice
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEQvsCONC (TRA-047)
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Helicobacter Pylori
MeSH Terms: interventions — Amoxicillin; Metronidazole; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequential treatment: (Active Comparator)
  Interventions: Drug: PPI, amoxicillin, metronidazole and clarithromycin
- Concomitant treatment (Experimental)
  Interventions: Drug: PPI, amoxicillin, metronidazole and clarithromycin

INTERVENTIONS:
Drug: PPI, amoxicillin, metronidazole and clarithromycin — Dual therapy for 5 days: PPI and 1g amoxicillin every 12h. After dual therapy continue with a triple therapy for 5 days: PPI, 1g amoxicillin, 500 mg metronidazole and 500 mg clarithromycin every 12h.
  Arms: Sequential treatment:
Drug: PPI, amoxicillin, metronidazole and clarithromycin — Quadruple therapy for ten days:PPI, 1g amoxicillin, 500 mg metronidazole and 500 mg clarithromycin every 12h
  Arms: Concomitant treatment

SUMMARY:
Helicobacter pylori is the main cause of chronic gastritis, peptic ulcer and gastric tumors (adenocarcinoma and lymphoma). The cure of the H. pylori infection prevents recurrence of duodenal and gastric ulcer and improves dyspepsia in a significant proportion of cases, so it is cost-effective.

Eradication therapy has changed over time. The usually recommended pattern in the consensus conferences has traditionally been triple therapy, composed by the combination of 2 antibiotics (clarithromycin plus amoxicillin or metronidazole) and a proton pump inhibitor (PPI) for 7-14 days. Recent meta-analyses have that the current global eradication rate after standard triple therapy is less than 80%. Several European studies have found even lower eradication rates, with 35-40% of cases resulting in treatment failure. Treatment failure leads to a second treatment and a new diagnostic test to confirm eradication.

DETAILED DESCRIPTION:
Justification of the study:

One of the latest therapeutic innovations is sequential therapy, introduced in Italy by Zullo et al. The drug delivery strategy involves a 5-day induction phase with dual therapy (a PPI every 12 hours and amoxicillin 1g every 12 hours), followed immediately by triple therapy for 5 days with a PPI every 12 hours, metronidazole 500 mg every 12 hours and clarithromycin 500 mg every 12 hours. Sequential therapy has proved more effectiveness than standard triple therapy for seven and ten days. In order to assess the efficacy of this new treatment in our area, over the past year we conducted a multicentre observational pilot study in routine clinical practice conditions in patients infected with H. pylori and with indications for eradication. 139 patients from 6 different centres were included. Excellent treatment compliance and minimal side effects, similar to those described with triple therapy, were shown. The results confirm similar efficacy to that obtained in previous studies and an eradication rate significantly higher than that obtained with classic triple therapy in our area.

Several previous studies have shown excellent efficacy of quadruple therapy with a PPI, amoxicillin, clarithromycin and metronidazole, administering "concomitantly" the same drugs as those of sequential therapy, but only for 5-7 days. Several studies have found a higher eradication rate of this "concomitant" therapy as compared with classic triple therapy. The results of a randomized study in which sequential and concomitant therapy were compared have recently been reported in the American Congress of Gastroenterology. Eradication and adverse events rates were similar with both treatments. This data suggest that the "sequentially"administration of these drugs probably complicated unnecessarily the treatment.

Therefore it is necessary to make a controlled clinical trial to directly compare "sequential" versus "concomitant" therapy. The results of this study will conclude which should be the first line treatment for H. pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion of patients with dyspepsia or peptic gastroduodenal ulcer for whom eradication treatment is indicated.
* Requirement of confirmation of the diagnosis of H. pylori infection by at least one positive test out of the following: breath test, histology, rapid urease test or culture.

Exclusion Criteria:

* Age less than 18 years.
* Advanced chronic disease or any other pathology that prevents attending controls and follow up.
* Allergy to any of the antibiotics in the treatment.
* Previous gastric surgery
* Pregnancy and lactation.
* History of alcohol or drug abuse.
* Previous eradication treatment.
* Consumption of antibiotics or bismuth salts during the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
"Intention to treat" eradication rates | One year
  "Intention-to-treat" eradication of infection.

SECONDARY OUTCOMES:
"Per protocol" Eradication rate | One year
  "Per protocol" eradication of infection.
Compliance | One year
  Treatment compliance
Adverse events | One year
  Adverse events
Clinical and demographic variables | One year
  Age Sex Smoking habits Comorbidity (diabetes mellitus, arterial hypertension, ischemic heart disease, dyslipidemia, others) Indication for eradication (peptic ulcer vs. uninvestigated or functional dyspepsia) Initial diagnostic test for H. pylori infection.

CONTACTS AND LOCATIONS:
Overall Officials: Javier P. Gisbert, Physician Doctor, Principal Investigator — Digestive Service, Hospital Universitario de La Princesa
Locations (11):
- Spain (11):
  - Hospital del Mar, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital de Cabueñes, Gijón
  - Hospital San Jorge, Huesca
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Costa del Sol, Málaga
  - Hospital de Sabadell, Sabadell
  - Hospital Universitario de Valme, Seville
  - Hospital Mútua de Terrassa, Terrassa
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital Clínico Universitario "Lozano Blesa", Zaragoza

REFERENCES:
- [Background] Forbes GM, Glaser ME, Cullen DJ, Warren JR, Christiansen KJ, Marshall BJ, Collins BJ. Duodenal ulcer treated with Helicobacter pylori eradication: seven-year follow-up. Lancet. 1994 Jan 29;343(8892):258-60. doi: 10.1016/s0140-6736(94)91111-8. PMID 7905095
- [Background] Howden CW, Hunt RH. Guidelines for the management of Helicobacter pylori infection. Ad Hoc Committee on Practice Parameters of the American College of Gastroenterology. Am J Gastroenterol. 1998 Dec;93(12):2330-8. doi: 10.1111/j.1572-0241.1998.00684.x. No abstract available. PMID 9860388
- [Background] Laheij RJ, Rossum LG, Jansen JB, Straatman H, Verbeek AL. Evaluation of treatment regimens to cure Helicobacter pylori infection--a meta-analysis. Aliment Pharmacol Ther. 1999 Jul;13(7):857-64. doi: 10.1046/j.1365-2036.1999.00542.x. PMID 10383518
- [Background] Calvet X, Ducons J, Bujanda L, Bory F, Montserrat A, Gisbert JP; Hp Study Group of the Asociacion Espanola de Gastroenterologia. Seven versus ten days of rabeprazole triple therapy for Helicobacter pylori eradication: a multicenter randomized trial. Am J Gastroenterol. 2005 Aug;100(8):1696-701. doi: 10.1111/j.1572-0241.2005.50019.x. PMID 16086704
- [Background] Calvet X, Garcia N, Lopez T, Gisbert JP, Gene E, Roque M. A meta-analysis of short versus long therapy with a proton pump inhibitor, clarithromycin and either metronidazole or amoxycillin for treating Helicobacter pylori infection. Aliment Pharmacol Ther. 2000 May;14(5):603-9. doi: 10.1046/j.1365-2036.2000.00744.x. PMID 10792124
- [Background] Gene E, Calvet X, Azagra R, Gisbert JP. Triple vs. quadruple therapy for treating Helicobacter pylori infection: a meta-analysis. Aliment Pharmacol Ther. 2003 May 1;17(9):1137-43. doi: 10.1046/j.1365-2036.2003.01566.x. PMID 12752350
- [Background] Zullo A, Rinaldi V, Winn S, Meddi P, Lionetti R, Hassan C, Ripani C, Tomaselli G, Attili AF. A new highly effective short-term therapy schedule for Helicobacter pylori eradication. Aliment Pharmacol Ther. 2000 Jun;14(6):715-8. doi: 10.1046/j.1365-2036.2000.00766.x. PMID 10848654
- [Background] Zullo A, Vaira D, Vakil N, Hassan C, Gatta L, Ricci C, De Francesco V, Menegatti M, Tampieri A, Perna F, Rinaldi V, Perri F, Papadia C, Fornari F, Pilati S, Mete LS, Merla A, Poti R, Marinone G, Savioli A, Campo SM, Faleo D, Ierardi E, Miglioli M, Morini S. High eradication rates of Helicobacter pylori with a new sequential treatment. Aliment Pharmacol Ther. 2003 Mar 1;17(5):719-26. doi: 10.1046/j.1365-2036.2003.01461.x. PMID 12641522
- [Background] Zullo A, Gatta L, De Francesco V, Hassan C, Ricci C, Bernabucci V, Cavina M, Ierardi E, Morini S, Vaira D. High rate of Helicobacter pylori eradication with sequential therapy in elderly patients with peptic ulcer: a prospective controlled study. Aliment Pharmacol Ther. 2005 Jun 15;21(12):1419-24. doi: 10.1111/j.1365-2036.2005.02519.x. PMID 15948808
- [Background] Francavilla R, Lionetti E, Castellaneta SP, Magista AM, Boscarelli G, Piscitelli D, Amoruso A, Di Leo A, Miniello VL, Francavilla A, Cavallo L, Ierardi E. Improved efficacy of 10-Day sequential treatment for Helicobacter pylori eradication in children: a randomized trial. Gastroenterology. 2005 Nov;129(5):1414-9. doi: 10.1053/j.gastro.2005.09.007. PMID 16285942
- [Background] Scaccianoce G, Hassan C, Panarese A, Piglionica D, Morini S, Zullo A. Helicobacter pylori eradication with either 7-day or 10-day triple therapies, and with a 10-day sequential regimen. Can J Gastroenterol. 2006 Feb;20(2):113-7. doi: 10.1155/2006/258768. PMID 16482238
- [Background] De Francesco V, Zullo A, Margiotta M, Marangi S, Burattini O, Berloco P, Russo F, Barone M, Di Leo A, Minenna MF, Stoppino V, Morini S, Panella C, Francavilla A, Ierardi E. Sequential treatment for Helicobacter pylori does not share the risk factors of triple therapy failure. Aliment Pharmacol Ther. 2004 Feb 15;19(4):407-14. doi: 10.1046/j.1365-2036.2004.01818.x. PMID 14871280
- [Background] Vaira D, Zullo A, Vakil N, Gatta L, Ricci C, Perna F, Hassan C, Bernabucci V, Tampieri A, Morini S. Sequential therapy versus standard triple-drug therapy for Helicobacter pylori eradication: a randomized trial. Ann Intern Med. 2007 Apr 17;146(8):556-63. doi: 10.7326/0003-4819-146-8-200704170-00006. PMID 17438314
- [Background] De Francesco V, Zullo A, Hassan C, Faleo D, Ierardi E, Panella C, Morini S. Two new treatment regimens for Helicobacter pylori eradication: a randomised study. Dig Liver Dis. 2001 Nov;33(8):676-9. doi: 10.1016/s1590-8658(01)80044-x. PMID 11785713
- [Background] Zullo A, De Francesco V, Hassan C, Morini S, Vaira D. The sequential therapy regimen for Helicobacter pylori eradication: a pooled-data analysis. Gut. 2007 Oct;56(10):1353-7. doi: 10.1136/gut.2007.125658. Epub 2007 Jun 12. PMID 17566020
- [Background] Sanchez-Delgado J, Calvet X, Bujanda L, Gisbert JP, Tito L, Castro M. Ten-day sequential treatment for Helicobacter pylori eradication in clinical practice. Am J Gastroenterol. 2008 Sep;103(9):2220-3. doi: 10.1111/j.1572-0241.2008.01924.x. Epub 2008 Jun 28. PMID 18564109
- [Background] Unge P. Review of Helicobacter pylori eradication regimens. Scand J Gastroenterol Suppl. 1996;215:74-81. PMID 8722388
- [Background] Sykora J, Siala K, Varvarovska J, Pazdiora P, Pomahacova R, Huml M. Epidemiology of Helicobacter pylori infection in asymptomatic children: a prospective population-based study from the Czech Republic. Application of a monoclonal-based antigen-in-stool enzyme immunoassay. Helicobacter. 2009 Aug;14(4):286-97. doi: 10.1111/j.1523-5378.2009.00689.x. PMID 19674133
- [Background] Vakil N. H. pylori treatment: new wine in old bottles? Am J Gastroenterol. 2009 Jan;104(1):26-30. doi: 10.1038/ajg.2008.91. PMID 19098845
- [Background] Graham DY, Lu H, Yamaoka Y. Therapy for Helicobacter pylori infection can be improved: sequential therapy and beyond. Drugs. 2008;68(6):725-36. doi: 10.2165/00003495-200868060-00001. PMID 18416582
- [Background] Graham DY, Lu H. Is there a role for sequential in sequential anti-H. pylori therapy? Gastroenterology. 2006 May;130(6):1930-1; author reply 1931. doi: 10.1053/j.gastro.2006.03.037. No abstract available. PMID 16697763
- [Background] Calvet X, Tito L, Comet R, Garcia N, Campo R, Brullet E. Four-day, twice daily, quadruple therapy with amoxicillin, clarithromycin, tinidazole and omeprazole to cure Helicobacter pylori infection: a pilot study. Helicobacter. 2000 Mar;5(1):52-6. doi: 10.1046/j.1523-5378.2000.00007.x. PMID 10672052
- [Background] Catalano F, Branciforte G, Catanzaro R, Cipolla R, Bentivegna C, Brogna A. Helicobacter pylori-positive duodenal ulcer: three-day antibiotic eradication regimen. Aliment Pharmacol Ther. 2000 Oct;14(10):1329-34. doi: 10.1046/j.1365-2036.2000.00839.x. PMID 11012478
- [Background] Gisbert JP, Marcos S, Gisbert JL, Pajares JM. High efficacy of ranitidine bismuth citrate, amoxicillin, clarithromycin and metronidazole twice daily for only five days in Helicobacter pylori Eradication. Helicobacter. 2001 Jun;6(2):157-62. doi: 10.1046/j.1523-5378.2001.00023.x. PMID 11422472
- [Background] Nagahara A, Miwa H, Ogawa K, Kurosawa A, Ohkura R, Iida N, Sato N. Addition of metronidazole to rabeprazole-amoxicillin-clarithromycin regimen for Helicobacter pylori infection provides an excellent cure rate with five-day therapy. Helicobacter. 2000 Jun;5(2):88-93. doi: 10.1046/j.1523-5378.2000.00013.x. PMID 10849057
- [Background] Nagahara A, Miwa H, Yamada T, Kurosawa A, Ohkura R, Sato N. Five-day proton pump inhibitor-based quadruple therapy regimen is more effective than 7-day triple therapy regimen for Helicobacter pylori infection. Aliment Pharmacol Ther. 2001 Mar;15(3):417-21. doi: 10.1046/j.1365-2036.2001.00929.x. PMID 11207518
- [Background] Neville PM, Everett S, Langworthy H, Tompkins D, Mapstone NP, Axon AT, Moayyedi P. The optimal antibiotic combination in a 5-day Helicobacter pylori eradication regimen. Aliment Pharmacol Ther. 1999 Apr;13(4):497-501. doi: 10.1046/j.1365-2036.1999.00493.x. PMID 10215734
- [Background] Okada M, Oki K, Shirotani T, Seo M, Okabe N, Maeda K, Nishimura H, Ohkuma K, Oda K. A new quadruple therapy for the eradication of Helicobacter pylori. Effect of pretreatment with omeprazole on the cure rate. J Gastroenterol. 1998 Oct;33(5):640-5. doi: 10.1007/s005350050150. PMID 9773927
- [Background] Okada M, Nishimura H, Kawashima M, Okabe N, Maeda K, Seo M, Ohkuma K, Takata T. A new quadruple therapy for Helicobacter pylori: influence of resistant strains on treatment outcome. Aliment Pharmacol Ther. 1999 Jun;13(6):769-74. doi: 10.1046/j.1365-2036.1999.00551.x. PMID 10383506
- [Background] Treiber G, Ammon S, Schneider E, Klotz U. Amoxicillin/metronidazole/omeprazole/clarithromycin: a new, short quadruple therapy for Helicobacter pylori eradication. Helicobacter. 1998 Mar;3(1):54-8. doi: 10.1046/j.1523-5378.1998.08019.x. PMID 9546119
- [Background] Treiber G, Wittig J, Ammon S, Walker S, van Doorn LJ, Klotz U. Clinical outcome and influencing factors of a new short-term quadruple therapy for Helicobacter pylori eradication: a randomized controlled trial (MACLOR study). Arch Intern Med. 2002 Jan 28;162(2):153-60. doi: 10.1001/archinte.162.2.153. PMID 11802748
- [Background] Essa AS, Kramer JR, Graham DY, Treiber G. Meta-analysis: four-drug, three-antibiotic, non-bismuth-containing "concomitant therapy" versus triple therapy for Helicobacter pylori eradication. Helicobacter. 2009 Apr;14(2):109-18. doi: 10.1111/j.1523-5378.2009.00671.x. PMID 19298338
- [Background] Wu DC, Hsu PI, Wu JY, Opekun AR, Kuo CH, Wu IC, Wang SS, Chen A, Hung WC, Graham DY. Sequential and concomitant therapy with four drugs is equally effective for eradication of H pylori infection. Clin Gastroenterol Hepatol. 2010 Jan;8(1):36-41.e1. doi: 10.1016/j.cgh.2009.09.030. Epub 2009 Oct 3. PMID 19804842
- [Derived] McNicholl AG, Marin AC, Molina-Infante J, Castro M, Barrio J, Ducons J, Calvet X, de la Coba C, Montoro M, Bory F, Perez-Aisa A, Forne M, Gisbert JP; Participant Centres. Randomised clinical trial comparing sequential and concomitant therapies for Helicobacter pylori eradication in routine clinical practice. Gut. 2014 Feb;63(2):244-9. doi: 10.1136/gutjnl-2013-304820. Epub 2013 May 11. PMID 23665990